CLINICAL TRIAL: NCT04512846
Title: Comparison of Efficacy in Stereotactic Body Radiation Therapy (SBRT) of Large Hepatocellular Carcinoma (5-10 cm) With or Without Transcatheter Arterial Chemoembolization (TACE)
Brief Title: Comparison of Efficacy in SBRT of Large HCC With or Without TACE
Status: Recruiting | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: large HCC with/without TACE
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-03

CONDITIONS: Large HCC Patients; Stereotactic Body Radiation Therapy; Transcatheter Arterial Chemoembolization
Keywords: CyberKnife; SBRT; large HCC; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CK-SBRT with TACE group: The hepatocellular carcinoma patients (5-10cm）who received SBRT with TACE.
- CK-SBRT group: The hepatocellular carcinoma patients (5-10cm）who received SBRT alone.

SUMMARY:
The study aims to compare efficacy and adverse reactions of large hepatocellular carcinoma participants (5-10cm) who receive stereotactic body radiation therapy with or without transcatheter arterial chemoembolization.The investigators will optimize the combined treatment schedule of SBRT for hepatocellular carcinoma participants by comparing overall survival rates, progression-free survival rates and local control and adverse reaction occurrence rates in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* primary HCC diagnosed by a surgeon and/or radiologist and oncologist according to the international guidelines for the management of HCC or by pathology
* single lesion and longest tumor diameter were 5-10cm;
* CP-A or B classification;
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* distances between tumor and normal organs (esophagus, stomach, duodenum, bowel) are more than 5 mm
* unsuitable for other therapies, such as patients with heart disease, uncontrolled diabetes, uncontrolled hypertension, etc.
* rejecting other therapies such as resection, liver transplantation, etc.
* platelet count≥50 × 109/L, white blood count≥1.5 × 109/L;
* patients infected with hepatitis B virus who are treated with adefovir or entecavir; patients infected with hepatitis C virus whose HCV DNA are negative.

Exclusion Criteria:

* tumor thrombus;
* lymph node involvement;
* extrahepatic metastasis.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The large HCC patients who receive SBRT with or without TACE.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | From date of randomization until the date of death from any cause, assessed up to 36 months
  OS is calculated starting from the date of SBRT to the date of the final follow-up or demise of the patients.
Progression-free survival time | From date of randomization until the date of disease progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS is estimated starting from the date of SBRT to the date of disease progression or patient death.
Local control time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  LC is defined starting from the date of SBRT to the date of treated-lesion progression or patient death.

SECONDARY OUTCOMES:
Radiation-induced liver injury rates | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
Adverse reaction | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing 302 hospital, Beijing, China

REFERENCES:
- [Result] Su TS, Lu HZ, Cheng T, Zhou Y, Huang Y, Gao YC, Tang MY, Jiang HY, Lian ZP, Hou EC, Liang P. Long-term survival analysis in combined transarterial embolization and stereotactic body radiation therapy versus stereotactic body radiation monotherapy for unresectable hepatocellular carcinoma >5 cm. BMC Cancer. 2016 Nov 3;16(1):834. doi: 10.1186/s12885-016-2894-9. PMID 27809890
- [Result] Wong TC, Chiang CL, Lee AS, Lee VH, Yeung CS, Ho CH, Cheung TT, Ng KK, Chok SH, Chan AC, Dai WC, Wong FC, Luk MY, Leung TW, Lo CM. Better survival after stereotactic body radiation therapy following transarterial chemoembolization in nonresectable hepatocellular carcinoma: A propensity score matched analysis. Surg Oncol. 2019 Mar;28:228-235. doi: 10.1016/j.suronc.2019.01.006. Epub 2019 Jan 29. PMID 30851906
- [Result] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569